CLINICAL TRIAL: NCT04980950
Title: "The Impact of Enteral Immunonutrition on Gut Microbiota, Intestinal Permeability, and Inflammation of Intestines in Colorectal Cancer as Well as Gastric Cancer Patients - a Randomized Trials"
Brief Title: "The Impact of Immunonutrition on Gut Microbiota-related Aspects in Colorectal Cancer and Gastric Cancer Patients"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Karolina Kaźmierczak-Siedlecka, Karolina Kaźmierczak-Siedlecka (nutritionist, PhD), senior assistant, Department of Surgical Oncology, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MUG
Record Dates: First submitted 2021-04-21; First posted 2021-07-28 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Gastric Cancer; Colorectal Cancer
Keywords: gut microbiota; gut barrier integrity; enteral immunonutrition; gastric cancer; colorectal cancer
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- gastric cancer patients (immunonutrition) (Experimental): Experimental gastric cancer group will receive Impact Oral Nestlé Health Science/ Cubitan® Nutricia for 10 days.
  Interventions: Dietary Supplement: Impact Oral Nestlé Health Science, Cubitan® Nutricia, Nutridrink® Nutricia, Resource 2.0 Nestlé Health Science
- gastric cancer patients (standard nutrition) (Active Comparator): These patients will receive Nutridrink® Nutricia/ Resource 2.0 Nestlé Health Science for 10 days.
  Interventions: Dietary Supplement: Impact Oral Nestlé Health Science, Cubitan® Nutricia, Nutridrink® Nutricia, Resource 2.0 Nestlé Health Science
- colorectal cancer patients (immunonutrition) (Experimental): Experimental colorectal cancer group will receive Impact Oral Nestlé Health Science/ Cubitan® Nutricia for 10 days.
  Interventions: Dietary Supplement: Impact Oral Nestlé Health Science, Cubitan® Nutricia, Nutridrink® Nutricia, Resource 2.0 Nestlé Health Science
- colorectal cancer patients (standard nutrition) (Active Comparator): These patients will receive Nutridrink® Nutricia/ Resource 2.0 Nestlé Health Science for 10 days.
  Interventions: Dietary Supplement: Impact Oral Nestlé Health Science, Cubitan® Nutricia, Nutridrink® Nutricia, Resource 2.0 Nestlé Health Science

INTERVENTIONS:
Dietary Supplement: Impact Oral Nestlé Health Science, Cubitan® Nutricia, Nutridrink® Nutricia, Resource 2.0 Nestlé Health Science — Gastric and colorectal cancer patients will receive 1 bottle of immunonutrition or standard nutrition for 10 days. The aims of this study is to assess the effects of these immunonutrition on gut microbiota, intestinal permeability as well as inflammation of intestines in gastric and colorectal cancer patients.

SUMMARY:
Enteral immunomodulating nutrition modifies the gastrointestinal microbiota as well as improves the intestinal barrier integrity in patients with gastric and colorectal cancer in the perioperative period. As a consequence, it contributes to the reduction of the incidence of postoperative complications and diarrhea, which is a side effect of anti-cancer treatment often used preoperatively in this group of cancers.

ELIGIBILITY:
Inclusion Criteria:

* age >18 y.o.
* patients with gastric or colorectal cancer
* patients treated in Department of Surgical Oncology, Medical University of Gdańsk
* patients' agreement to take part in this study

Exclusion Criteria:

* age <18 y.o.
* other types of cancer than gastric/colorectal cancer
* the presence of inflammatory bowel disease
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
The impact of immunonutrition on gut microbiota in gastric and colorectal cancer patients. | at baseline and after 7 and 10 days
  The composition of gut microbiota (bacteria and fungi) will be assessed from stools. The amounts of bacteria/fungi will be presented using bioinformatics tools and there is no precisely described units (only the total number).

SECONDARY OUTCOMES:
The impact of immunonutrition on intestinal permeability in gastric and colorectal cancer patients. | at baseline and after 7 and 10 days
  The ratio lactulose/mannitol will be described to assess intestinal permeability. There is no units. Only ratio of two numbers.
The impact of immunonutrition on intestines in gastric and colorectal cancer patients. | at baseline and after 7 and 10 days
  The calprotecin will be assessed. The unit is μg/g.

IPD SHARING:
Plan to Share IPD: No